CLINICAL TRIAL: NCT00597857
Title: Prevention of PTSD With Early Hydrocortisone Treatment: Pilot
Brief Title: Prevention of Posttraumatic Stress Disorder (PTSD) With Early Hydrocortisone Treatment: Pilot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kent State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Douglas L. Delahanty, PhD, Kent State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 05-025; R34MH073014 (NIH)
Record Dates: First submitted 2008-01-10; First posted 2008-01-18 (Estimated); Last update posted 2009-01-28 (Estimated); Status verified 2009-01

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): receipt of a placebo pill for 16 days
  Interventions: Drug: placebo
- 2 (Active Comparator): oral pill of hydrocortisone (ranging from 20mg - 2.5mg) taken for 10 days with a taper for 6 days (based on Pitman et al, 2002).
  Interventions: Drug: Hydrocortisone

INTERVENTIONS:
Drug: Hydrocortisone — Participants will receive a tapering low-dose of hydrocortisone in pill form for 10 days, twice a day, after the trauma.
  Other Names: Cortisol; Cortef; Hydrocortone
  Arms: 2
Drug: placebo — receipt of a placebo pill for 16 days
  Arms: 1

SUMMARY:
People experience a wide range of outcomes following a traumatic event. Although rates differ depending on type of trauma, 20-60% of trauma victims may develop posttraumatic stress disorder (PTSD). However, not all trauma victims develop PTSD. Previous research has found that trauma victims who develop PTSD excrete lower levels of urinary cortisol immediately after a trauma than victims who do not develop PTSD. Other research has suggested that increasing levels of cortisol may protect against the development of PTSD in patients such as yourself- but this has not yet been examined. Cortisol is a naturally occurring hormone in your body, and the present study is designed to test whether increasing cortisol levels can protect against or decrease symptoms of PTSD. Participants in this study will be randomly assigned to one of two treatment groups. Participants will receive either hydrocortisone (20mg, twice per day) or a placebo (a sugar pill) for 10 days with a six-day taper. There is an equal chance of being in either treatment group, and neither the participant nor the experimenters will know which treatment was received (except in case of an emergency).

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is the fourth most common psychiatric disorder and is estimated to affect more than ten million American children and adults at some point in their lives. Although a number of pre-, peri-, and acute phase post-trauma variables (e.g., prior trauma history, subjective life threat, injury) have been shown to increase one's risk of developing PTSD, initial psychological reaction to a traumatic event is an imperfect predictor of subsequent diagnosis. In addition, early psychological interventions have generally proven ineffective, and in some cases, detrimental with regards to subsequent symptomatology. In light of this, researchers have recently begun to examine possible pharmacological interventions that could be administered in the acute phase of responding to trauma to prevent or reduce the severity of subsequent post-traumatic stress.

Biopsychological research has frequently (but not always) indicated that patients with PTSD excrete lower levels of cortisol than similarly-exposed trauma victims who do not develop PTSD. Further, recent research has shown that lower cortisol levels present soon after a trauma are associated with increased risk for developing PTSD symptoms. These results suggest that higher levels of cortisol during and immediately after a traumatic event may buffer the development of PTSD symptoms. In addition, preliminary findings have suggested that exogenously elevating patients' levels of cortisol during and immediately following trauma results in decreased incidence of PTSD. However, these data were collected on relatively small samples of trauma patients with confounding medical conditions (e.g., shock, cardiac surgery, or paralysis). A randomized controlled trial (RCT) is necessary to determine the efficacy of early cortisol administration at buffering the development of post-traumatic stress in a heterogeneous trauma sample.

Prior to conducting a large-scale RCT, it is necessary to pilot test the efficacy of early cortisol treatment at reducing or preventing PTSD symptoms in a representative sample of heterogeneous trauma victims. The proposed research is designed to examine the efficacy of hydrocortisone (commercially-available cortisol) in preventing post-traumatic stress in a small-scale, randomized, double-blind trial. More specifically, incidence of PTSD and comorbid disorders (i.e., mood, anxiety and substance abuse/dependence disorders), severity of symptoms, health-related quality of life, and hormonal correlates of distress will be prospectively examined in trauma victims who are randomly assigned to receive either a course of hydrocortisone or placebo within 12 hours of the traumatic event. As psychological and physiological reactions to trauma may develop over a number of months post-trauma, prospective follow-up will allow us to examine the efficacy of cortisol administration at reducing both early as well as delayed development of symptoms. The proposed research will provide pilot data and effect size estimates for a subsequent large-scale trial, should pilot results be promising.

Specific objectives of the proposed research include:

1. Examination of the effects of early (within 12 hours of trauma) cortisol administration on subsequent symptoms of PTSD in trauma victims. Specifically, victims admitted to the Level 1 trauma unit of a local hospital will be randomly assigned to receive double-blind, low-dose cortisol (20mg, twice daily: bid) or placebo for ten days plus a 6-day taper period. Symptoms of psychopathology will be measured at 1- and 3-months post-trauma. Secondary analyses will examine the effects of cortisol on disorders commonly comorbid with PTSD (i.e., anxiety, mood, and substance abuse/dependence disorders) and on health-related quality of life.
2. Examination of the extent to which early cortisol administration influences the relationship between preexisting and trauma-related factors and psychophysiological responses to trauma. In particular, as lifetime incidence of psychopathology, prior trauma exposure, and injury severity have been associated with increased risk for PTSD, we will examine whether this relationship is weakened in patients receiving the cortisol regimen. Due to budgetary constraints of the R34 mechanism and the exploratory nature of the proposed research, we will not be able to recruit enough participants to sufficiently examine this objective, and it is thus considered a secondary aim. However, results will be used to strengthen and guide the design of a subsequent R01 proposal.

ELIGIBILITY:
Inclusion Criteria:

* involved in a traumatic event and admitted to the level 1 trauma center within 12 hours after the trauma

Exclusion Criteria:

* Glasgow coma scale score of less than 14 (at the time that you speak to patient)
* Amnestic for the events during and immediately following the traumatic event
* Unable to understand consent procedure or current substance abuse
* Traumatic event occurred more than 12 hours before initial medication dose can be given (i.e., patient life-flight or transferred after significant time has passed).
* Allergy to cortisol.
* Pregnant or breast-feeding
* Traumatic event of potentially ongoing nature that the participant is likely to be re-exposed to during the study (e.g. domestic violence)
* Presence of injuries (e.g. pelvic or lower extremity fractures) requiring readmission for surgery 1-2 weeks later once swelling has diminished. Patients requiring such delayed operative procedures will be excluded.
* Presence of medical condition that contraindicates the administration of cortisol, including (but not necessarily limited to) peptic ulcers, Cushing's disease, hypothyroidism, current alcoholism or cirrhosis, hepatitis, diverticulitis, nonspecific ulcerative colitis, myasthenia gravis, seizure disorders, renal insufficiency, disorders of immunosuppression, current viral or bacterial infection, diabetes mellitus, history of myocardial infarction, or recipient of solid organ or bone marrow transplant.
* On a current corticosteroid regimen (inhaled, oral, or injection). This may include patients with asthma, multiple sclerosis, arthritis, allergic conditions, optic neuritis, or tuberculosis
* Corticosteroid use in the previous 6 months
* Current use of medications that may have potentially dangerous interactions with cortisol including other corticosteroids, any immunosuppressant medications, drugs affecting hepatic microsomal enzymes, cyclosporine, and anticholinesterase agents.
* Injuries requiring treatment with steroids (e.g., suspected spinal cord injury, cerebral edema).
* Patients must be able to take oral medications within 12 hours post-trauma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2005-06; Primary Completion 2009-08 (Estimated); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
Clinician-Administered PTSD Scale (CAPS) | one- and three-months post-trauma

CONTACTS AND LOCATIONS:
Overall Officials: Doulas L Delahanty, PhD, Principal Investigator — Kent State University
Locations (1):
- Akron City Hospital, Akron, Ohio, United States

REFERENCES:
- [Background] Delahanty DL, Raimonde AJ, Spoonster E. Initial posttraumatic urinary cortisol levels predict subsequent PTSD symptoms in motor vehicle accident victims. Biol Psychiatry. 2000 Nov 1;48(9):940-7. doi: 10.1016/s0006-3223(00)00896-9. PMID 11074232
- [Background] Delahanty, D.L., Royer, D.K., Spoonster, E., & Raimonde, A.J. (2003). Peritraumatic dissociation is inversely related to catecholamine levels in initial urine samples of motor vehicle accident victims. Journal of Trauma and Dissociation, 4, 65-80.
- [Background] Flesher MR, Delahanty DL, Raimonde AJ, Spoonster E. Amnesia, neuroendocrine levels and PTSD in motor vehicle accident victims. Brain Inj. 2001 Oct;15(10):879-89. doi: 10.1080/02699050110065682. PMID 11595084
- [Background] Delahanty DL, Raimonde AJ, Spoonster E, Cullado M. Injury severity, prior trauma history, urinary cortisol levels, and acute PTSD in motor vehicle accident victims. J Anxiety Disord. 2003;17(2):149-64. doi: 10.1016/s0887-6185(02)00185-8. PMID 12614659
- [Background] Delahanty DL, Bogart LM, Figler JL. Posttraumatic stress disorder symptoms, salivary cortisol, medication adherence, and CD4 levels in HIV-positive individuals. AIDS Care. 2004 Feb;16(2):247-60. doi: 10.1080/09540120410001641084. PMID 14676029
- [Background] Pitman RK, Sanders KM, Zusman RM, Healy AR, Cheema F, Lasko NB, Cahill L, Orr SP. Pilot study of secondary prevention of posttraumatic stress disorder with propranolol. Biol Psychiatry. 2002 Jan 15;51(2):189-92. doi: 10.1016/s0006-3223(01)01279-3. PMID 11822998
- [Background] Schelling G, Kilger E, Roozendaal B, de Quervain DJ, Briegel J, Dagge A, Rothenhausler HB, Krauseneck T, Nollert G, Kapfhammer HP. Stress doses of hydrocortisone, traumatic memories, and symptoms of posttraumatic stress disorder in patients after cardiac surgery: a randomized study. Biol Psychiatry. 2004 Mar 15;55(6):627-33. doi: 10.1016/j.biopsych.2003.09.014. PMID 15013832
- [Background] Schelling G, Briegel J, Roozendaal B, Stoll C, Rothenhausler HB, Kapfhammer HP. The effect of stress doses of hydrocortisone during septic shock on posttraumatic stress disorder in survivors. Biol Psychiatry. 2001 Dec 15;50(12):978-85. doi: 10.1016/s0006-3223(01)01270-7. PMID 11750894